CLINICAL TRIAL: NCT00004066
Title: A Phase II Trial of Gemcitabine and Docetaxel in Patients With Unresectable Leiomyosarcoma
Brief Title: Gemcitabine, Docetaxel, and Filgrastim in Treating Patients With Recurrent or Persistent Leiomyosarcoma or Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-027; P30CA008748 (NIH); MSKCC-99027; NCI-G99-1576
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Ovarian Cancer; Sarcoma; Small Intestine Cancer
Keywords: adult leiomyosarcoma; recurrent adult soft tissue sarcoma; small intestine leiomyosarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; uterine leiomyosarcoma; ovarian sarcoma; recurrent small intestine cancer; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Ovarian Neoplasms; Sarcoma; Leiomyosarcoma | interventions — Filgrastim; Docetaxel; Gemcitabine

INTERVENTIONS:
Biological: filgrastim
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine, docetaxel, and filgrastim in treating patients who have recurrent or persistent leiomyosarcoma or soft tissue sarcoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the activity of gemcitabine plus docetaxel administered with filgrastim (G-CSF) support, in terms of disease response, in patients with recurrent or persistent unresectable leiomyosarcoma or other soft tissue sarcoma.
* Determine the tolerability of this regimen in these patients.
* Correlate response with tumor expression of the apoptosis-regulating proteins bax, bcl-2, and survivin in these patients.

OUTLINE: Patients are stratified according to prior radiotherapy to the pelvis (yes vs no).

Patients receive gemcitabine IV over 90 minutes on days 1 and 8 followed by docetaxel IV over 1 hour on day 8 and filgrastim (G-CSF) subcutaneously on days 9-15. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with a partial response may receive 2 additional courses of therapy.

Patients are followed every 3 months for 1 year or until disease progression.

PROJECTED ACCRUAL: A total of 38-82 patients (19-43 with uterine leiomyosarcoma and 19-39 with other soft tissue sarcoma) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed leiomyosarcoma (LMS) or other soft tissue sarcoma

  * No gastrointestinal stromal tumors, chondrosarcoma, Kaposi's sarcoma, Ewing's sarcoma, osteosarcoma, or mesotheliomas
* Recurrent or progressive disease defined as an increase in the size of any existing tumor (or the development of new tumors) that is not amenable to definitive surgical therapy
* No prior chemotherapy OR
* Failed no more than 2 prior chemotherapy regimens for LMS of the uterus or other soft tissue sarcoma
* Bidimensionally measurable disease by physical examination or medical imaging techniques

  * Ascites and pleural effusions are not considered measurable disease
* No uncontrolled CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No active or uncontrolled infection
* No other prior malignancy except non-metastatic squamous cell or basal cell skin cancer or non-invasive carcinoma in situ of the cervix
* No history of grade 3 or 4 peripheral neuropathy
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy
* No prior gemcitabine or docetaxel

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 6 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 1999-06; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Hensley ML, Maki R, Venkatraman E, Geller G, Lovegren M, Aghajanian C, Sabbatini P, Tong W, Barakat R, Spriggs DR. Gemcitabine and docetaxel in patients with unresectable leiomyosarcoma: results of a phase II trial. J Clin Oncol. 2002 Jun 15;20(12):2824-31. doi: 10.1200/JCO.2002.11.050. PMID 12065559